CLINICAL TRIAL: NCT05269472
Title: Trigeminal Evoked Responses to Improve Rhizotomy
Brief Title: Trigeminal Neuralgia Electrophysiology
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NSU-2022-30582
Record Dates: First submitted 2022-02-24; First posted 2022-03-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trigeminal Electrophysiology
  Interventions: Procedure: Trigeminal Electrophysiology
- Controls

INTERVENTIONS:
Procedure: Trigeminal Electrophysiology — This study will pilot and test the feasibility of introducing electrophysiology into the routine rhizotomy procedure by including trigeminal somatosensory evoked potentials (TSEPs) and recording from electrodes at the level of the ganglion.
  Groups: Trigeminal Electrophysiology

SUMMARY:
The study intervention is to perform standard somatosensory evoked responses limited to the face during rhizotomy procedures of the gasserian ganglion (trigeminal ganglion) for the treatment of trigeminal neuralgia. The evoked responses will be measured at two locations before and after the clinical rhizotomy including: the standard contralateral scalp (EEG) and at the gasserian ganglion through an FDA-approved recording electrode.

ELIGIBILITY:
Inclusion Criteria (TGN):

* Adults of 18 years or older
* Scheduled to undergo percutaneous rhizotomy for facial pain

Exclusion Criteria (TGN):

* Facial pain of unclear origin (i.e. not clearly TGN pain)
* Rhizotomy procedure canceled

Inclusion Criteria (Healthy controls)

* Adults of 18 years or older

Exclusion Criteria (Healthy Controls)

* Diagnosis or history of facial pain such as TMD or TGN
* History of migraine
* History of any functional pain disorder: fibromyalgia, IBS, CRPS
* Recent chronic pain (within last month)
* Unwilling to participate for two hours in lab
* Current acute pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults of 18 years or older who are scheduled to undergo percutaneous rhizotomy for facial pain
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility of measuring trigeminal somatosensory evoked potentials to improve personalized mapping during percutaneous rhizotomy | 3 years
  percentage of consented participants who complete the study

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States